CLINICAL TRIAL: NCT04665193
Title: An Approach to Screening for SARS-CoV-2 at YVR: UBC-PHC-WestJet-YVR COVID-19 Screening Study
Brief Title: An Approach to Screening for COVID-19 at Vancouver Airport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Airport Authority (Unknown); WestJet Airlines (Unknown); Providence Health & Services (Other); KLM Royal Dutch Airlines (Unknown)
Responsible Party: Principal Investigator, Don Sin, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H20-03225
Record Dates: First submitted 2020-12-08; First posted 2020-12-11 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Asymptomatic Condition; Healthy
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abbott Panbio test device (Experimental): WestJet passengers departing from YVR screened for COVID-19 using Abbott Panbio test device
  Interventions: Diagnostic Test: Rapid Antigen Test

INTERVENTIONS:
Diagnostic Test: Rapid Antigen Test — Antigen Technology Lab-based test and Point of care test
  Other Names: Abbott Rapid Diagnostics Panbio Covid-19 Ag Rapid Test Device (Nasopharyngeal)

SUMMARY:
The primary objective of this pilot study is to determine the feasibility and effectiveness of a COVID-19 screening program for passengers departing from YVR. This research study is conducted by The University of British Columbia (UBC) and Providence Health Care, sponsored by WestJet and Vancouver Airport Authority. The experimental study investigates point-of-care rapid test device for detecting SARS-CoV-2, the virus responsible for COVID-19. The study is investigating a method of rapid-testing for COVID-19 and will help inform the safest and most efficient way of testing departing passengers prior to security screening at Vancouver International Airport (YVR). This study is also evaluating a new passenger management system.

DETAILED DESCRIPTION:
Summary of the Research Proposal

Purpose:

The purpose of this pilot study is to determine the feasibility and effectiveness of a COVID-19 screening program at YVR for WestJet and KLM passengers.

Hypothesis:

SARS-CoV-2 infection can be effectively screened using point-of-care rapid antigen assays.

Justification:

Passengers are required to wear masks and physically distance while traveling by air. However, the majority of general public is still worried about the potential risk of contracting COVID-19 on airplanes, especially during long flights. We need to develop methods and strategies to quickly screen for SARS-CoV-2 infection, prior to boarding flights.

Objectives:

1. To develop and deploy a management algorithm for COVID-19 screening at YVR that will involve the use of point-of-care rapid test device.
2. To evaluate the acceptability of such screening algorithm and determine the costs of deploying the program.

Research Design:

Study Population: Working in collaboration with WestJet and KLM we will invite all passengers meeting Inclusion/Exclusion on outbound flights from YVR Airport to participate in this study.

Phase 1: We will work with YVR and WestJet to enroll 200 subjects into the study. For this initial phase we are looking to determine the rate of positivity in the cohort. This initial phase is needed to evaluate the feasibility of this pilot program and to refine the initial management algorithm. Health Canada-approved Panbio Covid-19 Ag Rapid Test Device by Abbott Rapid Diagnostics (approved for Lab-based test and Point of care test on 2020-10-05) will be uses in Phase 1.

Phase 2: Strategies for achieving higher-throughput will be determined after completion of Phase 1. In phase 2, we will continue to work with YVR and WestJet, with the addition of KLM, to enroll 700 subjects into the study. Phase 2 will further assess the efficiency of our COVID-19 screening and passenger management algorithm.

The study is purposefully designed to be as minimally invasive to the passengers' travel plan as possible. The Study Plans for Phase 1 and Phase 2 are detailed below.

Statistical Analysis:

• When we aggregate the data for analysis, we will use basic statistics to determine mean, variance, standard deviation, and positivity rate...etc.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

1. The subject must be between 19 and 80 years of age.
2. The subject must be a resident of B.C.
3. The subject must have a ticket to board a WestJet flight departing from Vancouver International Airport (YVR).
4. Have a minimum of 75 minutes of free time prior to the scheduled flight's departure.

Phase 2 Inclusion Criteria:

1. Subject has access to accommodation in Canada for safe-isolation as per public health guidelines
2. Between the ages of 13 - 90
3. Travelling on any WestJet or KLM flight
4. Have a minimum of 70 minutes (if travelling within Canada) or 90 minutes (if travelling International) of free time prior to the schedule flight's departure

   -----------------------------------

   Exclusion Criteria:
   * Subjects who have previously tested positive for COVID-19 within the past 90 days
   * Subjects who cannot provide written informed consent

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
COVID-19 status | 15 minutes
  positive or negative screening result

CONTACTS AND LOCATIONS:
Overall Officials: Don Sin, MD, Principal Investigator — University of British Columbia; Marc Romney, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver International Airport, WestJet Domestic Terminal, Level 3, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04665193/Prot_002.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04665193/ICF_003.pdf